CLINICAL TRIAL: NCT07299981
Title: Quantitative Net Water Uptake as a Predictor of Functional Outcomes After Intravenous Thrombolysis in Acute Ischemic Stroke International Multicenter Observational Retrospective Study
Status: Not yet recruiting | Type: Observational
Sponsor: Sigmund Freud PrivatUniversitat (Other)
Responsible Party: Sponsor
Other Study IDs: 17803148
Record Dates: First submitted 2025-12-10; First posted 2025-12-23 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with ischemic stroke receiving IVT
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: No Interventions — Not applicable as this is an observational, retrospective study.

SUMMARY:
While the effectiveness of intravenous thrombolysis (IVT) decreases over time, patients show considerable variability in how quickly their ischemic core progresses. Quantitative net water uptake (NWU) has emerged as a biomarker indicating blood-brain barrier disruption and may better reflect the "tissue clock" than time alone. Low NWU is associated with favorable outcomes, whereas high NWU predicts poor outcomes and futile recanalization. The study aims to determine whether NWU measured on initial non-contrast CT is a treatment effect modifier for the IVT therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke treated with intravenous thrombolysis
* Imaging with non-contrast cranial CT on admission
* Follow-up imaging with non-contrast cranial CT or MRI 12-24 hours after IVT
* Final Infarct volume > 5ml
* ASPECTS available

Exclusion Criteria:

* Known use of oral anticoagulation (OAC) on admission
* Preexisting ischemic infarction on admission non-contrast cranial CT
* Patients with large vessel occlusion AIS who underwent mechanical thrombectomy
* Low imaging quality precluding radiological measurements
* Severe white matter lesions precluding radiological measurements
* No ASPECTS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged over 18 years with acute ischemic stroke, symptom onset within 24 hours prior to admission and treatment in one of the stroke units of the participating institutions between 2018 and 2025 treated using IVT and fullfilling inclusion criteria
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with functional independence (modified Rankin Scale score 0-1) | at 90 days
  Functional independence defined as a modified Rankin Scale (mRS) score of 0-1 assessed at 90 days.

SECONDARY OUTCOMES:
Number of participants with symptomatic intracerebral hemorrhage | at 24 hours
  Symptomatic intracerebral hemorrhage (sICH) as defined by the European Cooperative Acute Stroke Study (ECASS) III criteria (i.e., an ICH associated with an increase of ≥4 points on the NIHSS or death where intracranial hemorrhage is the predominant cause of neurological deterioration).
Number of participants with intracerebral hemorrhage on follow-up brain imaging | at 24 hours
  Intracerebral hemorrhage detected on follow-up brain imaging performed within 24 hours after treatment.
Mortality | at 90 days

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results after deidentification
Supporting Information: Study Protocol, SAP
Access Criteria: Data that support the findings of this study will be available from the corresponding author after academic board review and upon reasonable request